CLINICAL TRIAL: NCT01254227
Title: Phase II, Open-label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of Deferasirox in Combination With Deferoxamine Followed by Deferasirox Monotherapy in Patients With Severe Cardiac Iron Overload Due to Chronic Blood Transfusion (HYPERION)
Brief Title: Efficacy and Safety of Deferasirox in Combination With Deferoxamine Followed by Deferasirox Monotherapy in Severe Cardiac Iron Overload
Acronym: HYPERION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2214; 2010-021062-29 (EudraCT Number)
Record Dates: First submitted 2010-09-21; First posted 2010-12-06 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Iron Overload
Keywords: Cardiac iron overload,; deferasirox,; deferoxamine
MeSH Terms: interventions — Deferasirox; Deferoxamine

ARMS (1):
- Deferasirox (Experimental): Deferoxamine combination followed by Deferasirox monotherapy
  Interventions: Drug: Deferasirox and Deferoxamine

INTERVENTIONS:
Drug: Deferasirox and Deferoxamine

SUMMARY:
This study will evaluate the efficacy and safety of deferasirox in combination with deferoxamine followed be deferasirox monotherapy in patients with severe iron overload due to chronic blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with β-thalassemia major or Diamond-Blackfan anemia (DBA) or congenital sideroblastic anemia on chronic transfusion therapy
* Myocardial T2* value that is ≥ 5 and < 10 ms
* Left ventricular ejection fraction (LVEF) ≥ 56% as determined by Magnetic resonance imaging (MRI)
* Liver Iron Concentration (LIC) ≥ 7 mg Fe /g dw as determined by R2 MRI.
* Lifetime history of at least 50 units of red blood cell transfusions, and must be receiving at least ≥ 8 units/yr of red blood cell transfusions
* Serum ferritin ≥ 1000 ng/mL

Exclusion Criteria:

* Patients with clinical symptoms of cardiac dysfunction (shortness of breath at rest or exertion, orthopnea, exercise intolerance, lower extremity edema, arrhythmias)
* Patients unable to undergo study assessments including MRI
* Patients with serum creatinine greater than Upper limit of normal ULN)range or with significant proteinuria as indicated by a urinary protein/creatinine ratio (UPCR) ≥1.0 mg/mg in a non-first void urine sample at baseline.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Cairo, Egypt
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Patra - RIO, GR
- Italy (3):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Aydinok Y, Kattamis A, Cappellini MD, El-Beshlawy A, Origa R, Elalfy M, Kilinc Y, Perrotta S, Karakas Z, Viprakasit V, Habr D, Constantinovici N, Shen J, Porter JB; HYPERION Investigators. Effects of deferasirox-deferoxamine on myocardial and liver iron in patients with severe transfusional iron overload. Blood. 2015 Jun 18;125(25):3868-77. doi: 10.1182/blood-2014-07-586677. Epub 2015 May 1. PMID 25934475
- See also: link to the results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 centers in 8 countries.
Pre-assignment Details: A total 60 participants were enrolled in the study of which 34 completed the study.
Groups:
- All Participants: Participants received an initial combined dose of Deferasirox (DFX) 20 Milligrams per Kilogram per day (mg/kg/day) every day and Deferoxamine (DFO) 40 mg/kg/day (DFO: 5 days/week for at least 8 hours/day). Deferasirox was increased to 30 mg/kg/day every day at Month 1 Further dose increases upto 40 mg/kg/day every day at Month 6 visit. Participants could be switched from the Deferasirox - Deferoxamine (DFX - DFO) combination to Deferasirox monotherapy at the highest tolerable dose (30-40 mg/kg/day) at any time point after 6 months.
Period: Overall Study
Arm/Group | All Participants
Started | 60
Completion of 12 Months | 39
Completion of 24 Months | 34
Completed | 34
Not Completed | 26
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 5
Not completed — Abnormal test procedure result | 5
Not completed — Administrative problems | 2
Not completed — Death | 1
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received an initial combined dose of Deferasirox (DFX) 20 mg/kg/day every day and Deferoxamine (DFO) 40 mg/kg/day (DFO: 5 days/week for at least 8 hours/day). Deferasirox was increased to 30 mg/kg/day every day at Month 1 Further dose increases upto 40 mg/kg/day every day at Month 6 visit. Participants could be switched from the Deferasirox - Deferoxamine (DFX - DFO) combination to Deferasirox monotherapy at the highest tolerable dose (30-40 mg/kg/day) at any time point after 6 months.
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Iron Content From Baseline to Month 12
Description: Cardiac T2* is the most sensitive and reproducible test in detecting myocardial iron load. A cardiac T2* value of <10 ms is defined as severe cardiac iron overload. Participants who do not have baseline T2* or do not have any post-baseline T2* are excluded from the analysis.
Time Frame: From Baseline to Month 12
Population: The Full Analysis Set includes all participants to whom study treatment had assigned. Participants were considered evaluable for the efficacy endpoint if they had received at least one dose of study treatment and had baseline and a post baseline assessment prior to or on the time of the assessment of the corresponding efficacy endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 60
ratio | 1.09 [1.04 to 1.15]

2. Secondary Outcome: Percentage of Participants With T2*>=10 ms and at Least 10% Relative Increase From Baseline at Month 6, 12, 18 and 24
Description: The number of evaluable participants at each visit were used as the denominator for the calculation of proportion at each visit.
Time Frame: From the Months 6, 12, 18 and 24
Population: The Full Analysis Set includes all participants to whom study treatment had assigned. Participants were considered evaluable for the efficacy endpoint if they had received at least one dose of study treatment and had baseline and a post baseline assessment prior to or on the time of the assessment of the corresponding efficacy endpoint. Here, "Number of participants analyzed" included all participants who were evaluable for the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 44
percentage of participants
  Month 6: number analyzed (Participants) | 6
  Month 6 | 12.50 [5.86 to 24.70]
  Month12: number analyzed (Participants) | 10
  Month12 | 19.23 [10.80 to 31.90]
  Month 18: number analyzed (Participants) | 11
  Month 18 | 33.33 [19.75 to 50.39]
  Month 24: number analyzed (Participants) | 17
  Month 24 | 47.22 [31.99 to 62.99]

3. Secondary Outcome: Change in Cardiac Iron Content From Baseline to Month 6,18 and 24
Description: The change in cardiac iron content was calculated as ratio of Cardiac T2* at different time points; the efficacy endpoint analyses were performed on the Full Analysis Set (FAS).
Time Frame: From Baseline to Months 6, 18 and 24
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 60
ratio
  Month 6: number analyzed (Participants) | 48
  Month 6 | 1.02 [0.98 to 1.07]
  Month 18: number analyzed (Participants) | 33
  Month 18 | 1.17 [1.08 to 1.28]
  Month 24: number analyzed (Participants) | 36
  Month 24 | 1.30 [1.17 to 1.44]

4. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) From Baseline to Month 6, 12, 18 and 24
Description: Magnetic resonance imaging (MRI)-measured cardiac T2* and cardiac function reflected by left and right ventricle ejection fraction. A standardized MRI protocol for T2* acquisition technique will be used in the centers. Images will be reviewed centrally by an expert MRI reader.
Time Frame: From the Months 6, 12, 18 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | All Participants
Number analyzed (Participants) | 60
Percent Ejection Fraction
  Baseline | 66.5 (5.32)
  Month 6: number analyzed (Participants) | 48
  Month 6 | 0.1 (4.62)
  Month 12: number analyzed (Participants) | 45
  Month 12 | -0.2 (4.84)
  Month 18: number analyzed (Participants) | 33
  Month 18 | 0.6 (7.04)
  Month 24: number analyzed (Participants) | 36
  Month 24 | 0.9 (5.98)

5. Secondary Outcome: Change in Right Ventricular Ejection Fraction (RVEF) From Baseline to Month 6, 12, 18 and 24
Description: as for outcome 4
Time Frame: From the Months 6, 12, 18 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | All Participants
Number analyzed (Participants) | 60
Percent Ejection Fraction
  Baseline | 67.1 (5.55)
  Month 6: number analyzed (Participants) | 47
  Month 6 | -1.2 (5.35)
  Month 12: number analyzed (Participants) | 45
  Month 12 | -1.6 (4.40)
  Month 18: number analyzed (Participants) | 33
  Month 18 | -2.1 (6.10)
  Month 24: number analyzed (Participants) | 36
  Month 24 | -1.4 (4.25)

6. Secondary Outcome: Time to Achieve From Baseline (FAS) of at Least 10% at Month 24
Description: Time from date of start of study treatment to date when first achieving T2* ≥ 10 ms (but at least 10% relative increase from baseline) was summarized using the reverse Kaplan-Meier estimates (1 - Kaplan-Meier estimates) for the FAS.
Time Frame: At 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: milliseconds/ms
Arm/Group | All Participants
Number analyzed (Participants) | 60
milliseconds/ms | 722.0 [520.0 to NA] — NA: It was not estimable.

7. Secondary Outcome: Cardiac Iron Concentration Levels From Baseline and at Month 6, 12, 18 and 24
Description: Cardiac iron concentration (mg Fe/g dw) was quantified using the formula (cardiac iron concentration (mg Fe/g dw) = 45 * T2* (ms) ^ (-1.22) and analyzed over time.
Time Frame: From the Baseline, Month 6, 12, 18 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | All Participants
Number analyzed (Participants) | 60
mg Fe/g dw
  Baseline | 4.18 (1.045)
  Month 6: number analyzed (Participants) | 48
  Month 6 | 4.31 (1.442)
  Month 12: number analyzed (Participants) | 46
  Month 12 | 3.93 (1.429)
  Month 18: number analyzed (Participants) | 33
  Month 18 | 3.51 (1.348)
  Month 24: number analyzed (Participants) | 36
  Month 24 | 3.14 (1.381)

ADVERSE EVENTS:
Time Frame: All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit, up to 24 months with 28 days of Follow up
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 17/60
Other Adverse Events (participants affected / at risk) | 52/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=60)
Anaemia (Blood and lymphatic system disorders) | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abscess neck (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Calcium deficiency (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=60)
Thrombocytosis (Blood and lymphatic system disorders) | 2
Atrioventricular block first degree (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Conductive deafness (Ear and labyrinth disorders) | 2
Deafness bilateral (Ear and labyrinth disorders) | 2
Deafness neurosensory (Ear and labyrinth disorders) | 3
Eustachian tube dysfunction (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Toothache (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 4
Influenza like illness (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 14
Acute tonsillitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 4
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 4
Tooth abscess (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 10
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2
Traumatic arthritis (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 5
Cardiac murmur (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 2
Electrocardiogram T wave amplitude decreased (Investigations) | 3
Electrocardiogram T wave inversion (Investigations) | 4
Urine protein/creatinine ratio increased (Investigations) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes